CLINICAL TRIAL: NCT01395615
Title: Utility Measurement Study for Patients With Chronic Lymphocytic Leukaemia
Brief Title: An Observational Study on The Health Related Quality of Life in Patients With Chronic Lymphocytic Leukaemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22686
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will assess the health related quality of life (HQRL) profiles of patients with chronic lymphocytic leukaemia. Using health assessment questionnaires, data will be collected from patients currently receiving therapy and from those who have finished therapy and have undergone an assessment of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with chronic lymphocytic leukaemia
* Patients receiving 1st line therapy
* Patients receiving 2nd line therapy. This will include patients who previously have responded well to 1st line therapy (relapse was >12 months after finishing the 1st line therapy) and are receiving the same therapy again
* Within the past three months, patients whose treatment has been stopped after 2-3 cycles of 1st or 2nd line therapy and who have not received any further therapies
* Patients receiving their 3rd, 4th, 5th or 6th cycle of 1st or 2nd line therapy
* Patients who have completed therapy, are considered stable and are between 3-12 months post therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* Clinically significant disorder (other than chronic lymphocytic leukaemia and chronic lymphocytic comorbidities) or any other condition, including alcohol or drug abuse, which may interfere with study participation or affect study conclusions
* Mental disability or significant mental illness, legal incapacity or limited legal capacity
* Current high degree of comorbid burden that might affect the accuracy of the quality of life data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lymphocytic leukaemia
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Quality of life: EuroQol Group EQ-5D questionnaire | 18 months
Quality of life: European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire | 18 months
Quality of life: EORTC QLQ-CLL16 (chronic lymphocytic leukaemia) questionnaire | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United Kingdom (4):
  - Bournemouth
  - Leeds
  - London
  - Taunton